CLINICAL TRIAL: NCT04323293
Title: Pain Modulation - Experimental Assessments Using Different Modalities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Schweinhardt Petra (Other)
Responsible Party: Sponsor-Investigator, Schweinhardt Petra, Head of Research Department of Chiropractic Medicine, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pain modulation assessments
Record Dates: First submitted 2020-03-11; First posted 2020-03-26 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Low Back Pain; Compare Pain Modulation Assessments in Pain-free Cohorts
Keywords: low back pain; temporal summation of pain; conditioned pain modulation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Participants (pain-free controls or patients with low back pain) will undergo either only one intervention (cold water bath) or two interventions in randomized order (cold water bath, water bath of neutral temperature as SHAM condition).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are unaware of the hypothesis. Outcomes assessors in subprojects are blind to the type of the water bath.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPM - Cold Water Bath (Experimental)
  Interventions: Other: Cold Water Bath
- CPM - SHAM (Sham Comparator)
  Interventions: Other: Neutral Water Bath

INTERVENTIONS:
Other: Cold Water Bath — immersion of the hand for 2-5min in 2-10°C water
  Arms: CPM - Cold Water Bath
Other: Neutral Water Bath — immersion of the hand for 2-5min in 32±2°C water
  Arms: CPM - SHAM

SUMMARY:
The goal of this study is to investigate how different painful stimuli are processed and modulated in the nervous system. In various pain conditions, including low back pain, often no specific source can be identified as the cause of the pain. Scientific findings point towards a possible involvement of sensitization processes in the central nervous system (spinal cord and brain) that can contribute to the development and persistence of chronic pain. There is a need for reliable and well established experimental methods to better investigate and understand these processes. Frequently used methods comprise the application of thermal, mechanical or electrical stimulations. These modalities are processed in different parts of the nervous system, each allowing its own conclusions. This can be an advantage, but it also poses a challenge regarding comparability and generalizability of obtained results.

This study aims to apply and compare various experimental methods in people without and people with low back pain and shed light on the methodological differences. In the future, this could enable better identification and characterization of sensitization processes in the nervous system and build the basis for individually adapted, mechanism-targeted treatments with better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* German or English proficiency
* Informed consent
* primary pain complaint localized between the 12th rib and the gluteal fold
* low back pain for more than one week
* low back pain clinically not attributable to "red flags" (including infection, trauma, fractures, inflammatory)

Exclusion Criteria:

* unable to give informed consent (e.g. due to language problems)
* any neurological condition
* any major medical or psychiatric condition (e.g. severe heart disease, diabetes, autoimmune disorders, major depressive disorder), any chronic pain condition other than low back pain
* pregnancy
* Radiating pain below knee level (radicular pain)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 705 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Temporal Summation of Pain (TSP) | 1-4 weeks
  TSP is measured as the change in perceived pain over time in response to repetitive noxious stimulation. In this study, a series of stimulations will be applied using different modalities (pressure, superficial mechanical, heat or electrical stimuli). Participants will be asked to report the perceived pain in response to the stimulations on an 11-point numerical rating scale (0: no pain, 10: most intense pain) or a visual analogue scale (VAS). VAS will be anchored with 0 ("no sensation"), 40 ("just painful," defined as the pain threshold), and 100 ("most intense pain tolerable"). Reflex parameters (thresholds in milliampere (mA); amplitude in μV) will be recorded at start and end of the series. Differences in read-outs (pain ratings, reflex thresholds or reflex amplitudes) at the start of the series compared to the end of the series or the slope of the pain ratings over the series will serve as TSP measures. Greater differences (end-start) or steeper slopes represent a greater TSP.
Conditioned Pain Modulation (CPM) | 1-4 weeks
  CPM measures the modulation of a noxious test stimulus by another noxious conditioning stimulus applied at a remote body region. In this study, test stimuli of different modalities (pressure, superficial mechanical, heat or electrical stimuli) will be applied at different body regions before and after or before, during and after a cold water bath or neutral water bath (hand immersion) as conditioning stimulus. Changes in test stimuli read-outs (during-before or after-before) will serve as CPM measure. Negative changes represent inhibitory, positive changes facilitatory CPM effects. For all test stimuli read-outs, CPM effects will be expressed as percentage changes.
  Test stimuli read-outs include: pain ratings (numerical rating scale or VAS, anchors see TSP outcome); perception thresholds (in kg for pressure, millinewton for superficial mechanical, °C for heat and mA for electrical stimuli); pain thresholds; reflex parameters (thresholds in mA and/or amplitudes).
CPM effect on TSP | 1-4 weeks
  Changes in TSP in response to the intervention (conditioning stimulus: cold water bath or SHAM).

SECONDARY OUTCOMES:
Pressure sensory and pain sensitivity | 1-4 weeks
  Pressure sensitivity will be assessed by for example perception and pain thresholds measured in kg/cm^2. Low thresholds reflect greater sensitivity.
Mechanical sensory and pain sensitivity | 1-4 weeks
  Mechanical (superficial) sensitivity will be assessed by for example perception and pain thresholds measured in millinewton. Low thresholds reflect greater sensitivity.
Heat sensory and pain sensitivity | 1-4 weeks
  Heat sensitivity will be assessed by for example perception and pain thresholds measured in °C. Low thresholds reflect greater sensitivity.
Electrical sensory and pain sensitivity | 1-4 weeks
  Electrical sensitivity will be assessed by for example perception, pain and reflex thresholds measured in milliampere. Low thresholds reflect greater sensitivity.
Pain Catastrophizing | 1-4 weeks
  Pain catastrophizing will be assessed using questionnaires as for example the Pain Catastrophizing Scale (0-52; higher score meaning more catastrophizing).
Fear of pain | 1-4 weeks
  Fear of pain will be assessed using questionnaires as for example the Fear Avoidance Belief Questionnaire (0-96) or the Tampa Scale of Kinesiophobia (17-69; higher scores meaning greater fear of pain).
Anxiety | 1-4 weeks
  Anxiety will be assessed using questionnaires as for example the Spielberger's State and Trait Anxiety Inventory (20-80; higher scores meaning greater anxiety).
  depression (e.g., Becks Depression Inventory(0-63); higher scores meaning greater level of depression).
Depression | 1-4 weeks
  Depression will be assessed using questionnaires as for example the Becks Depression Inventory (0-63; higher scores meaning greater level of depression).
Pain duration | 1-4 weeks
  Low back pain patients will be asked to indicate the duration of their clinical pain in months/years.
Spatial pain extent | 1-4 weeks
  Low back pain patients will be asked to complete pain drawings indicating painful body regions. The painful body area will be calculated as percentage of the whole body area. Higher percentages represent more widespread pain.
Somatic symptoms | 1-4 weeks
  Additional questionnaires complementing the psychological construct "pain catastrophizing" are implemented in selected subprojects of the study, e.g., the "Somatic Symptom Scale - 8" (higher score meaning higher somatic symptom burden).

CONTACTS AND LOCATIONS:
Overall Officials: Petra Schweinhardt, PhD, Principal Investigator — Integrative Spinal Research, Department of Chiropractic Medicine, Balgrist University Hospital, University of Zurich
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland